CLINICAL TRIAL: NCT02842450
Title: Study of Photographs of Interest in Training to Obtain Good Reproducibility of the Diagnosis of Perianal Lesions of Crohn's Disease Inspection in Internal Gastroenterology
Acronym: PhotoCrohn
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PhotoCrohn
Record Dates: First submitted 2016-07-13; First posted 2016-07-22 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Crohn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- training with typical definitions established + photos: A broad group of experts (19 proctology and a dermatologist) will be contacted to choose two typical images of LAP (superficial ulceration, deep ulceration ...). 12 photos lesion initially selected by experts.
  Interventions: Device: Photos + definitions
- Training only with definitions: Interns will receive typical definitions of LAP stages
  Interventions: Other: definitions only

INTERVENTIONS:
Device: Photos + definitions — A broad group of experts (19 proctology and a dermatologist) will be contacted to choose two typical images of LAP (superficial ulceration, deep ulceration ...). 12 photos lesion initially selected by experts.
  Groups: training with typical definitions established + photos
Other: definitions only
  Groups: Training only with definitions

SUMMARY:
The diagnosis of LAP (lesions Ano-perineal) requires the inspection, palpation, anoscopy and possibly additional examinations including endoscopy and imaging; any of these steps of the diagnosis can only be replaced by another.

In the absence of data in the literature on the evaluation of specific LAP Crohn inspection, Clemence Horaist et al established definitions of these lesions inspection with the help of an expert group, then evaluated the diagnostic agreement LAP these definitions in the same group from a selection of photographs. Definitions ulceration, fistula, inflammatory external os, erythema and abscess had an acceptable agreement diagnosis (kappa> 0.70)

The LAP is a predictor of severe Crohn's disease, hepato any gastroenterologist it is appropriate that recognizes and adopts adequate care, this care has been a consensus in 2014. The interns Hepato gastroenterology must learn during their training to know the terminology of LAP Crohn inspection and to recognize so considered acceptable by experts.

DETAILED DESCRIPTION:
Study Objectives:

In this context, the investigators work is to show that training giving the consensus definitions of Crohn's lesions on inspection and typical images of these lesions is effective to enable students to achieve a level of diagnosis of these lesions acceptable to experts (ideally not significantly different from that of the experts). Assuming alternates, we will identify difficult diagnosis of lesions for students to find the most appropriate teaching method

Inclusion criteria: all Gastroenterology Hepato-house of France (including overseas territories)

Methodology:

non-interventional multicentre prospective study

February 2015 to July 2015

Statistical analysis: Clinical Research Centre of the coordinating center. Quantitative variables are expressed by their mean, standard deviations, their minimum and maximum values as appropriate. The variables will be expressed in numbers and percentages.

Development of the study:

* A broad group of experts (19 proctology and a dermatologist) will be contacted to choose two typical images of LAP (superficial ulceration, deep ulceration ...) from a selection of photos and give their opinions about fistula definition proposal. (Photos used does not identify patients, they have just typical lesions of LAP)

Typical pictures chosen by the experts will be integrated into the training material issued after 1 internal questionnaire. This support will appear on one page and resume the definitions established by experts with or without the typical pictures.

* Internal Gastroenterology France (about 470 domestic total) will be contacted by email, their department heads have been told that work.
* Internal will inform their characteristics:

  * Internal details: name, email address
  * Year boarding.
  * boarding area.
  * Validation IUD (inter-university degree) 1st / 2nd year of proctology.
  * Conducting an internal internship in a proctology service?
  * Participation in specific courses on the LAP?
  * buddy Training on LAP?
* Sending a first questionnaire to internal Google Drive: description pictures of LAP (12 photos lesion initially selected by experts) using checkboxes. Eg ulceration: YES / NO / DO NOT KNOW (Figure 1). The Google Drive platform enables automatic input results in a Microsoft Excel database.
* Draw (using a randomization list EXCEL based on the random function of EXCEL) of 2 groups:

  * Group A (training with typical definitions established + photos)
  * Group B (only definitions)
* Sending mail to the board of education, different depending on the group, the internal will have as long as they wish
* Sending a second questionnaire with pictures of different LAP those of the first questionnaire. Answers by checkboxes.
* Analysis: a schedule will each questionnaire with a weighting based on the primary / secondary diagnosis. A comparison of pre and post training scores will be performed. And this difference may be calculated between the two groups A and B. In addition, the difficult diagnosis of lesions will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Internal gastro enterology in France will be contacted by email, their department heads have been warned of this work

Exclusion Criteria:

* Internals who refuses the assessment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Internal gastro enterology in France (about 470 domestic total) will be contacted by email, their department heads have been warned of this work
Sampling Method: Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Assessment of the level (quality) of internal diagnosis of Perianal Lesions of Crohn's Disease Inspection | within 1 week after training
  Assessment the test scores after the training.
  The test conssite to evaluate whether training giving the consensus definitions of Crohn's lesions on inspection and typical images of these lesions is effective to enable students to achieve a good level of diagnosis of these lesions acceptable for experts (ideally not significantly different from that of the experts).

CONTACTS AND LOCATIONS:
Overall Officials: DE PARADES Vincent, MD, Principal Investigator — Groupe Hospitalier Paris Saint-Joseph (FRANCE)
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided